CLINICAL TRIAL: NCT05122351
Title: Comparative Study Between The Efficacy Of Quadratus Lumborum Block VS Conventional Analgesia In Patients Undergoing Open Inguinal Hernia Surgical Repair
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mamdouh Ahmed, Resident doctor at Anesthesia and ICU department, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-10-06
Record Dates: First submitted 2021-10-19; First posted 2021-11-16 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Analgesia in Patients With Open Inguinal Hernia Surgeries
MeSH Terms: interventions — Analgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of Bupivacaine infiltration at the Quadratus Lumborum muscle (Experimental): Patients will receive Quadratus Lumborum Block by infiltration of Bupivacaine as post operative analgesia in Open Inguinal Hernia surgery
  Interventions: Drug: Bupivacaine infiltration at the Quadratus Lumborum muscle Versus Paracetamol injection as analgesia in post operative Open Inguinal Hernia surgeries
- Group of paracetamol injection (Experimental): Patients will receive post operative 1 gm paracetamol injection as analgesia in Open Inguinal Hernia surgery
  Interventions: Drug: Bupivacaine infiltration at the Quadratus Lumborum muscle Versus Paracetamol injection as analgesia in post operative Open Inguinal Hernia surgeries

INTERVENTIONS:
Drug: Bupivacaine infiltration at the Quadratus Lumborum muscle Versus Paracetamol injection as analgesia in post operative Open Inguinal Hernia surgeries — Comparative Study Between The Efficacy Of Quadratus Lumborum Block VS Conventional Analgesia In Patients Undergoing Open Inguinal Hernia Surgical Repair

SUMMARY:
Analgesia In Patients Undergoing Open Inguinal Hernia Surgical Repair

DETAILED DESCRIPTION:
Comparative Study Between The Efficacy Of Quadratus Lumborum Block VS Conventional Analgesia In Patients Undergoing Open Inguinal Hernia Surgical Repair

ELIGIBILITY:
Inclusion Criteria:

* 50 patients with ASA grade I to II, posted for open inguinal hernia surgery, elective , 18 to 60 years old , will be included in double blinded randomized study.

Exclusion Criteria:

* Patient refusal
* Patient with significant neurological , psychiatric or neuromuscular disease.
* Pregnancy or lactating women.
* Suspected Coagulopathy .
* Morbid obesity.
* Known allergy to some medications .
* Septicaemia and local infection at the block site .
* Alcoholism .
* Drug abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Analgesia in Patients with Open Inguinal Hernia Surgeries | 6 months
  Comparative Study Between The Efficacy Of Quadratus Lumborum Block by Bupivacaine infiltration VS Conventional Analgesia by paracetamol injection In Patients Undergoing Open Inguinal Hernia Surgical Repair

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Joshi GP, Rawal N, Kehlet H; PROSPECT collaboration; Bonnet F, Camu F, Fischer HB, Neugebauer EA, Schug SA, Simanski CJ. Evidence-based management of postoperative pain in adults undergoing open inguinal hernia surgery. Br J Surg. 2012 Feb;99(2):168-85. doi: 10.1002/bjs.7660. Epub 2011 Sep 16. PMID 21928388
- [Background] Rab M, Ebmer And J, Dellon AL. Anatomic variability of the ilioinguinal and genitofemoral nerve: implications for the treatment of groin pain. Plast Reconstr Surg. 2001 Nov;108(6):1618-23. doi: 10.1097/00006534-200111000-00029. PMID 11711938
- [Background] Bulka CM, Shotwell MS, Gupta RK, Sandberg WS, Ehrenfeld JM. Regional anesthesia, time to hospital discharge, and in-hospital mortality: a propensity score matched analysis. Reg Anesth Pain Med. 2014 Sep-Oct;39(5):381-6. doi: 10.1097/AAP.0000000000000121. PMID 25025697